CLINICAL TRIAL: NCT04681703
Title: Efficacy of a Family Nurse-led Program on Accuracy of Blood Pressure Self-measurement: a Randomized Controlled Trial
Brief Title: Nurse-led Program Efficacy on Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti (Other)
Responsible Party: Principal Investigator, Giancarlo Cicolini, Principal Investigator, Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-19-2015
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Hypertension; Home Blood Pressure Measurement
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to usual care: a 1-h educational and training program conducted by the family nurse (FN) in a dedicated room of the ambulatory care centers. During the program, the nurse instructed patients on how to self-measure blood pressure (BP) using the BP self-measurement device and on the importance of adequate device maintenance. The intervention was carried out by the FN on a daily basis during outpatient visits of the participants to the general practitioner (GP).
  Interventions: Behavioral: Nurse-led program on accuracy of blood pressure self-measurement
- Conrol group (No Intervention): Management of hypertensive patients, usual care: verbal and written instructions during which the family nurse (FN) or general practitioner (GP) advised the patient to follow the recommendations regarding correct HBPM. A written summary of the recommendations was given to all participants by the GP or FN at the end of the training program.

INTERVENTIONS:
Behavioral: Nurse-led program on accuracy of blood pressure self-measurement — The training program was performed in accordance with current guidelines and consisted of a 1-h educational session led by one family nurse (FN) tasked with instruction of the patients. During the training program the FN emphasized that since morning and evening blood pressure (BP) values can widely differ, especially in patients taking medications, BP should be measured twice a day, in the morning and at evening, at specific fixed times (between 6:00 am and 9:00 am and between 6:00 pm and 9:00 pm) at least during the first week of monitoring. Thereafter, measurements can be taken before antihypertensive drugs are taken.
  Arms: Intervention group

SUMMARY:
The diagnosis and control of hypertension depend on accurate measurements of blood pressure (BP); alternative approaches to measuring BP, such as ambulatory blood pressure monitoring or home blood-pressure self-measurement (HBPM), are gaining increasing acceptance in the diagnosis of hypertension and the monitoring of hypertensive patients.To achieve accurate BP measurements at home, measurement guidelines must be closely followed. However, previous studies have shown that patient compliance is in most cases unsatisfactory.The study aims at evaluating the efficacy of a family nurse (FN)-led home blood pressure management (HBPM) training program in improving BP control based on a comparison with routine care and management.

DETAILED DESCRIPTION:
The quality of HBPM was found to be higher in patients who received some form of training in BP measurement from healthcare professionals than in patients who did not receive training. Although self-estimation of BP may be prone to error, this risk can be minimized through adequate patient education and training that includes simple but nonetheless important recommendations. However, unclear is whether specific training offered by nurses, who frequently have a close relationship with their hypertensive patients, could result higher patient adherence to HBPM recommendations. Therefore, we assume that a specifically tailored training program conducted by a family nurse (FN), when provided in addition to usual care, could improve patient adherence to HBPM recommendations.

Study design: single-blind, multicenter, randomized controlled trial.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of hypertension.
* Patients who visited one of two family practice offices located in Chieti or Pescara.
* Speaking and reading Italian.
* Having an active phone number and an email address.
* Providing a signed informed consent.

Exclusion Criteria:

* Mental illness.
* Cognitive impairments.
* Pregnancy.
* Institutionalization (nursing home).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change in percentage (%) of patients' adherence to the recommendations for corrrect home blood pressure measurement (HBPM) from baseline (T0) to 1 month (T1) | 1 month
  Response assessed using a structured questionnaire specifically designed to evaluate patients'adherence to current Italian guidelines on HBPM

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Cicolini, Principal Investigator — Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simonetti V, Comparcini D, Tomietto M, Pavone D, Flacco ME, Cicolini G. Effectiveness of a family nurse-led programme on accuracy of blood pressure self-measurement: A randomised controlled trial. J Clin Nurs. 2021 Aug;30(15-16):2409-2419. doi: 10.1111/jocn.15784. Epub 2021 Apr 19. PMID 33872417